CLINICAL TRIAL: NCT03619629
Title: Comparison of the Effects of Kinesio Taping and Mulligan's Mobilization With Movement on Balance, Muscle Strength and Flexibility in Healthy Ankles
Brief Title: Ankle Kinesio Taping vs Mulligan's Mobilization With Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Murat TOMRUK, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MullKT
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Kinesio-taping; Mulligan; Mobilization; balance; ankle
MeSH Terms: interventions — Athletic Tape; Movement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kinesio-taping (Experimental): Kinesiotape will be applied both ankles.
  Interventions: Other: Kinesio-tape
- Mulligan's mobilization with movement (Experimental): 'Posterolateral glide mobilization with movement' will be applied both ankles.
  Interventions: Other: Mulligan's mobilization with movement
- Sham Kinesio-taping (Sham Comparator): Sham kinesio-taping technique will be applied both ankles.
  Interventions: Other: Sham Kinesio-taping
- Sham Mulligan's mobilization with movement (Sham Comparator): Sham Mulligan's mobilization with movement will be applied both ankles.
  Interventions: Other: Sham Mulligan's mobilization with movement

INTERVENTIONS:
Other: Kinesio-tape — Kinesiotape will be applied both ankles as "Correction technique".
  Arms: Kinesio-taping
Other: Mulligan's mobilization with movement — 'Posterolateral glide mobilization with movement' will be applied 10 times to both ankles.
  Arms: Mulligan's mobilization with movement
Other: Sham Kinesio-taping — Sham Kinesio-taping technique will be applied both ankles.
  Arms: Sham Kinesio-taping
Other: Sham Mulligan's mobilization with movement — Sham Mulligan's mobilization with movement technique will be applied both ankles.
  Arms: Sham Mulligan's mobilization with movement

SUMMARY:
The aim of the study is to compare the effects of Kinesio taping and Mulligan's mobilization with movement technique on balance, muscle strength and flexibility in healthy ankles . Patients will randomly be divided into 4 groups: Kinesio taping (KT) group, sham Kinesio taping (SKT) group, Mulligan's mobilization with movement (MWM) group and sham mobilization with movement (SMWM) group . Kinesiotape will be applied both ankles as "Correction technique" in KT group, 'Posterolateral glide mobilization with movement' will be applied 10 times to both ankles in MWM group. The evaluations will be repeated after waiting 45 minutes to reveal the effects of Kinesio taping and Mulligan mobilization with movement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35
* Healthy individuals
* Able to read, write and understand Turkish
* willing and able to attend study

Exclusion Criteria:

* Any neurological, musculoskeletal or vascular disease in any of the lower extremity.
* Previous history of surgery in any of the lower extremity.
* Mental and cognitive disorders that would seriously affect cooperation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
change in balance | Before intervention and 45 minutes after the intervention
  Change in balance will be measured by using Biodex Balance System.

SECONDARY OUTCOMES:
change in muscle strength | Before intervention and 45 minutes after the intervention
  Change in muscle strength will be assessed by using hand-held dynamometer.
change in flexibility | Before intervention and 45 minutes after the intervention
  Change in flexibility will be assessed by weight-bearing lunge test
change in range of motion | Before intervention and 45 minutes after the intervention
  Change in range of motion will be assessed by using electronic gonyometer

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No